CLINICAL TRIAL: NCT05082688
Title: Exploratory Study Into Age-related Immunological Differences Related to Immunogenicity in Influenza Vaccination and Herpes Zoster Vaccination
Brief Title: Age Differences in Influenza and Herpes Zoster Vaccine Responses (INFLUENZA-SHINGRIX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL76061.091.20; 2020-005682-13 (EudraCT Number)
Record Dates: First submitted 2021-01-22; First posted 2021-10-19 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Influenza; Herpes Zoster
Keywords: Vaccination; Trained immunity; Immunosenescence; Inflammaging
MeSH Terms: conditions — Influenza, Human; Herpes Zoster | interventions — halofantrine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1: Young adults herpes zoster vaccination (Experimental): Young adults between 18 and 35 years old will receive the herpes zoster vaccine (Shingrix). 60 days later, they will receive a booster dose.
  Interventions: Biological: Herpes zoster vaccination (Shingrix, GSK)
- 2: Older adults herpes zoster vaccination (Experimental): Adults older than 60 years of age will receive the herpes zoster vaccine (Shingrix). 60 days later, they will receive a booster dose.
  Interventions: Biological: Herpes zoster vaccination (Shingrix, GSK)
- 3: Young adults influenza vaccination (Experimental): Young adults between 18 and 35 years old will receive the influenza vaccine (Fluarix Tetra).
  Interventions: Biological: Influenza Vaccine (Fluarix Tetra Northern Hemisphere 2021 or 2022, GSK)
- 4: Older adults influenza vaccination (Experimental): Adults older than 60 years of age will receive the influenza vaccine (Fluarix Tetra).
  Interventions: Biological: Influenza Vaccine (Fluarix Tetra Northern Hemisphere 2021 or 2022, GSK)
- 5: Young adults herpes zoster vaccination related placebo (Placebo Comparator): Young adults between 18 and 35 years old will receive the placebo injection (0.9% NaCl). 60 days later, they will receive another placebo.
  Interventions: Biological: Placebo
- 6: Young adults influenza vaccination related placebo (Placebo Comparator): Young adults between 18 and 35 years old will receive the placebo injection (0.9% NaCl).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes zoster vaccination (Shingrix, GSK) — Shingrix is an ASO1-adjuvanted herpes zoster vaccination used to prevent shingles and its associated complications in at-risk populations
  Arms: 1: Young adults herpes zoster vaccination; 2: Older adults herpes zoster vaccination
Biological: Influenza Vaccine (Fluarix Tetra Northern Hemisphere 2021 or 2022, GSK) — Fluarix Tetra is a quadrivalent inactivated influenza vaccine
  Arms: 3: Young adults influenza vaccination; 4: Older adults influenza vaccination
Biological: Placebo — 0.9% NaCl
  Arms: 5: Young adults herpes zoster vaccination related placebo; 6: Young adults influenza vaccination related placebo

SUMMARY:
Vaccines are used to prevent infectious diseases worldwide. Unfortunately, many vaccines, like the flu vaccine, are less effective in older adults.

This single-centre open label partially randomised, partially placebo-controlled trial evaluates the differences in immune response between young and older adults after vaccination with a quadrivalent inactivated influenza vaccine and an adjuvanted herpes zoster vaccination.

Exploring the underlying mechanisms between the differences in immunogenicity can provide important information for future vaccine development.

DETAILED DESCRIPTION:
Rationale: Vaccination of the older adults is often advised as they are a high-risk population; however, vaccine efficacy generally decreases with age. This is mainly due to a decrease in adaptive immune responses known as immunosenescence, which is a factor influencing the response to influenza vaccination. On the other hand, there are vaccines that show high efficacy (more than 95%) in older adults, one of the most effective being the AS01 adjuvanted herpes zoster vaccine, Shingrix. The differential immune pathways associated with vaccine responsiveness as well as the immune mechanisms by which adjuvants overcome immunosenescence remain poorly understood. Targeting key immune pathways could be a way to improve vaccine efficacy in older adults.

Objective: To explore immunological features between young and older adults after administration of an adjuvanted herpes zoster (Shingrix) or influenza unadjuvanted (Fluarix) vaccine that could explain differences in vaccine immunogenicity.

Study design: A single centre open label, randomised, and partially placebo-controlled trial Study population: Approximately 140 healthy adults, 80 of which are between 18-35 years old, the other 60 are 60+ years old.

Intervention: Two groups of young and elderly volunteers receive recombinant zoster vaccine (Shingrix), while two other groups will receive a quadrivalent influenza vaccine (Fluarix). Two groups of young volunteers will receive a placebo.

Main study parameter: To identify immune senescence-related differences contributing to vaccine immunogenicity

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years old OR age ≥60 years old
* Written informed consent

Exclusion Criteria:

* Known allergy to (components of) the influenza or herpes zoster vaccine
* Immunocompromised subjects and subjects with active malignancy within the last two years
* Previous herpes zoster vaccination in the last year
* Receipt of any vaccination 4 weeks prior to the start of the study or plans to receive any other vaccination in the first 2 months after inclusion
* Use of systemic immunomodulatory drugs:steroids, anti-inflammatory biological treatments (e.g. anti-cytokine monoclonal antibodies)
* Acute or active illness within two weeks prior to the start of the study
* Pregnant, breastfeeding or planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Changes in cytokine productions of PBMCs upon incubation with viral, bacterial, and fungal antigens | 2 months after influenza vaccination
  IL-6, TNF, IL-1b, IFNg cytokine concentrations will be measured.
Changes in cytokine productions of PBMCs upon incubation with viral, bacterial, and fungal antigens | 6 months after influenza vaccination
  IL-6, TNF, IL-1b, IFNg cytokine concentrations will be measured.
Changes in cytokine productions of PBMCs upon incubation with viral, bacterial, and fungal antigens | 2 months after the first dose of herpes zoster vaccination
  IL-6, TNF, IL-1b, IFNg cytokine concentrations will be measured.
Changes in cytokine productions of PBMCs upon incubation with viral, bacterial, and fungal antigens | 2 months after the second dose of herpes zoster vaccination
  IL-6, TNF, IL-1b, IFNg cytokine concentrations will be measured.
Changes in cytokine productions of PBMCs upon incubation with viral, bacterial, and fungal antigens | 6 months after the second dose of herpes zoster vaccination
  IL-6, TNF, IL-1b, IFNg cytokine concentrations will be measured.
Change in transcriptional profile of individual cells from PBMC population | 2 months after influenza vaccination
  Gene expression profile of PBMCs will be measured by single cell-RNA sequencing.
Change in transcriptional profile of individual cells from PBMC population | 6 months after influenza vaccination
  Gene expression profile of PBMCs will be measured by single cell-RNA sequencing.
Transcriptional profile of individual cells from PBMC population | 2 months after the first dose of herpes zoster vaccination
  Gene expression profile of PBMCs will be measured by single cell-RNA sequencing.
Transcriptional profile of individual cells from PBMC population | 2 months after the second dose of herpes zoster vaccination
  Gene expression profile of PBMCs will be measured by single cell-RNA sequencing.
Transcriptional profile of individual cells from PBMC population | 6 months after the second dose of herpes zoster vaccination
  Gene expression profile of PBMCs will be measured by single cell-RNA sequencing.

SECONDARY OUTCOMES:
Changes in the adaptive immune cell populations in blood | 2 months after influenza vaccination
  Ratio of adaptive immune cells (T and B cells) and their subtypes will be measured by FACS.
Changes in the adaptive immune cell populations in blood | 6 months after influenza vaccination
  Ratio of adaptive immune cells (T and B cells) and their subtypes will be measured by FACS.
Changes in the adaptive immune cell populations in blood | 2 months after the first dose of herpes zoster vaccination
  Ratio of adaptive immune cells (T and B cells) and their subtypes will be measured by FACS.
Changes in the adaptive immune cell populations in blood | 2 months after the second dose of herpes zoster vaccination
  Ratio of adaptive immune cells (T and B cells) and their subtypes will be measured by FACS.
Changes in the adaptive immune cell populations in blood | 6 months after the second dose of herpes zoster vaccination
  Ratio of adaptive immune cells (T and B cells) and their subtypes will be measured by FACS.
Baseline DNA methylation | Baseline (before vaccination)
  CpG methylation profile of PBMCs
Changes in B and T cell receptor repertoires | 2 months after influenza vaccination
  B and T cell receptors will be sequenced.
Changes in B and T cell receptor repertoires | 2 months after the first dose of herpes zoster vaccination
  B and T cell receptors will be sequenced.
Changes in B and T cell receptor repertoires | 2 months after the second dose of herpes zoster vaccination
  B and T cell receptors will be sequenced.
Changes in circulating protein concentrations | 2 months after influenza vaccination
  Concentrations of circulating inflammatory proteins, including TNF, IL-6, IL-8, CCL3, CCL4, CXCL9, CXCL10, CXCL11, will be measured by Olink.
Changes in circulating protein concentrations | 2 months after the first dose of herpes zoster vaccination
  Concentrations of circulating inflammatory proteins, including TNF, IL-6, IL-8, CCL3, CCL4, CXCL9, CXCL10, CXCL11, will be measured by Olink.
Changes in circulating protein concentrations | 2 months after the second dose of herpes zoster vaccination
  Concentrations of circulating inflammatory proteins, including TNF, IL-6, IL-8, CCL3, CCL4, CXCL9, CXCL10, CXCL11, will be measured by Olink.
Influenza vaccine-specific antibodies in the serum | 2 months after influenza vaccination
  HAI titers will be measured.
Shingles vaccine-specific antibody production in the serum | 2 months after the first herpes zoster vaccination
  Anti-gE titers will be measured.
Shingles vaccine-specific antibody production in serum | 2 months after the second herpes zoster vaccination
  Anti-gE titers will be measured.
Percentage of participants reporting local reactions | 7 days after influenza and herpes zoster vaccination
  Pain at the injection site, redness, and swelling
Percentage of participants reporting systemic events | 7 days after influenza and herpes zoster vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea
Changes in epigenetic markers in PBMCs | 2 months after influenza vaccination
  ATAC-sequencing will be performed to measure post transcriptional modifications (methylation, acetylation, etc) on histones.
Changes in epigenetic markers in PBMCs | 6 months after influenza vaccination
  ATAC-sequencing will be performed to measure post transcriptional modifications (methylation, acetylation, etc) on histones.
Changes in epigenetic markers in PBMCs | 2 months after the first herpes zoster vaccination
  ATAC-sequencing will be performed to measure post transcriptional modifications (methylation, acetylation, etc) on histones.
Changes in epigenetic markers in PBMCs | 2 months after the second herpes zoster vaccination
  ATAC-sequencing will be performed to measure post transcriptional modifications (methylation, acetylation, etc) on histones.
Changes in epigenetic markers in PBMCs | 6 months after the second herpes zoster vaccination
  ATAC-sequencing will be performed to measure post transcriptional modifications (methylation, acetylation, etc) on histones.
C-reactive protein in the serum | Baseline (before vaccination)
  Soluble C-reactive protein (CRP) concentrations will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap ten Oever, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Gelderland, Netherlands